CLINICAL TRIAL: NCT01112501
Title: SPECT/CT in the Diagnosis of Dementia
Acronym: DEMSPET
Status: Completed | Type: Observational
Sponsor: Kuopio University Hospital (Other)
Collaborators: University of Eastern Finland (Other)
Responsible Party: Esko Vanninen / Professor, Kuopio University Hospital
Other Study IDs: KUH5031339
Record Dates: First submitted 2010-04-27; First posted 2010-04-28 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Dementia
Keywords: Diagnosis; Dementia; Imaging
MeSH Terms: conditions — Dementia; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Aim of the study is to evaluate whether Tc-99m-ECD-SPECT/CT enhances early diagnosis of dementia in two specific patient groups: (1) patient with mild cognitive impairment, and (2) patient with possible symptoms and signs of frontotemporal dementia. Evaluation of SPECT/CT data is performed both by visual and quantitative voxel-based analyses (Statistical Parametric Mapping). The final diagnosis is based on up to four years clinical follow-up.

ELIGIBILITY:
Inclusion Criteria (one of these):

* healthy control
* mild cognitive impairment (recruited from a population based data)
* clinically suspected frontotemporal dementia (unset diagnosis)

Exclusion Criteria:

* unable to be scanned with SPECT/CT

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with possible/suspected early dementia
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2006-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Final diagnosis | 4 years
  (1) controls, (2) stable mild cognitive impairment (MCI), (3)MCI converted to Alzheimers's disease (AD), (4) frontotemporal dementia (FTD), suspected FTD converted to AD, (5) other final diagnoses

CONTACTS AND LOCATIONS:
Locations (1):
- Kuopio University Hospital, Kuopio, Finland